CLINICAL TRIAL: NCT05917730
Title: Clinical Trial for Promoting Emotional Regulation and Interpersonal Skills (MERITA) in Children and Adolescents Witnesses of Domestic Violence
Brief Title: Manual of Emotional Regulation and Interpersonal Abilities in Children and Adolescents Group Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Hospital Sant Joan de Deu (Other)
Responsible Party: Sponsor
Other Study IDs: PIC-90-20
Record Dates: First submitted 2023-03-02; First posted 2023-06-26 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Domestic Violence; Psychotherapy, Group; Witness
Keywords: Domestic Violence; Witness; Psychotherapy, Group; Clinical trial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: Emotional Regulation and Interpersonal Abilities group Therapy (MERITA).: 12 sessions of 75 minutes each and are carried out weekly. MERIT aims to improve emotional regulation, to cope with problems, promoting interpersonal skills and attachment security. Sessions will be lead by two psychologists with accredited experience in MERITA.
  Interventions: Behavioral: Emotional Regulation and Interpersonal Abilities group Therapy (MERITA)
- Control: Treatment As Usual: The treatment as usual provided in children and adolescents who witnesses DV is mainly individual psychotherapy.

INTERVENTIONS:
Behavioral: Emotional Regulation and Interpersonal Abilities group Therapy (MERITA) — Therapy sessions Block 1. Recognition and verbalization of emotions: Session 1: Presentation, framing, and beginning of identification and denomination of emotions. Session 2: Recognition and differentiation of emotions. Session 3 and 4: Effects of traumatic experiences.
  Block 2. Learning to manage emotions: Session 5: Managing unpleasant emotions, coping Abilities in body, mind, and behavior. Session 6: New coping skills, self-esteem. Session 7: New coping skills, self-care. Session 8: Skills for clear communication. Session 9: Assertiveness and reciprocity. Session 10: Save card and the good relations game/negotiation skills. Session 11: Social skills and confidence recovery. Session 12: Consolidation and farewell.
  Groups: Experimental: Emotional Regulation and Interpersonal Abilities group Therapy (MERITA).

SUMMARY:
Purpose:

Domestic violence (DV) is a mental health problem that affects children and adolescents. Widespread evidence suggests that witnessing DV has physical and mental health consequences. 19% of children and adolescents cared for in Children, and Youth Mental Health Centers in Catalonia declare having witnessed DV between their parents. However, there are low specialized therapeutic tools to intervene effectively. In this line, the research team of the current project adapted and manualized a group treatment designed to treat children and adolescents between 8 and 16 years old witnesses of DV on an outpatient basis called: 'Manual of Emotional Regulation and Interpersonal Abilities group Therapy - MERITA'. The treatment main aim is to improve the emotional regulation and interpersonal skills of children and adolescents who have witnessed DV. We carried out a pilot study of MERITA (Lacasa et al., 2016) where we obtained promising results. Now, we want to carry out this study to improve methodological limitations by increasing the sample size. We have added a waiting list for assigning patients in different arms (MERITA intervention vs. treatment as usual as control group), as well as we improved the assessment (pre, post, and follow-ups) using several scales with good psychometric properties.

Aims:

The aim of this trial is twofold: firstly, to assess the effectiveness of Emotional Regulation and Interpersonal Abilities group Therapy (MERITA) in children and adolescents who are witnesses of DV and treated at the Infant and dolescent mental health center (TAU); and secondly, to analyze the differences (MERITA vs only TAU) on traumatic, depressive and anxious symptomatology, emotional dysregulation, interpersonal difficulties, externalizing and internalizing symptoms, somatic complaints, prosocial behavior, attachment, and family functioning. Specifically, MERITA will be compared to TAU alone (post and 3-month follow-up).

Methods

Design:

Trail with two arms:

1. MERITA + TAU (intervention group)
2. TAU (control group)

Sample:

The necessary sample size to detect statistically significant differences between the groups has been calculated using the G*Power: with a minimum effect size (0.50), a significance level of 5% and a power of 80%. A minimum of 36 participants would be required.

DETAILED DESCRIPTION:
This clinical trial will be carried out with a group of children and adolescents who are witnesses of DV (between 8 and 16 years old). They will receive the MERITA treatment (together with TAU) and the other group will receive only TAU (control group).

The MERITA treatment consists of weekly 12 sessions of 75 minutes each. MERITA aims to improve emotional regulation and coping abilities, as well as promoting interpersonal skills and secure attachment.

After getting promising results from our previous pilot study of MERITA, the current project aims to validate, through a clinical trial with a control group, the MERIT treatment in minors who witness violence. To do this, children and adolescents who have undergone the MERIT will be compared with another group who receives other psychological and social approaches (treatment as usual), with other children and adolescents (same age and sex) who have only received treatment as usual.

The MERITA + TAU group and the TAU group will perform the following assessment: before treatment (baseline or pretreatment), after treatment (posttreatment), and at three months of follow-up. Specifically, the MERITA + TAU group will conduct two more assessments: at 6-month follow-up and one year of follow-up.

For ethical reasons, all patients will have the opportunity to use the MERITA treatment. Thus, the minors who were TAU group will go on to receive the MERITA treatment. It should be noted that these patients must have completed the 3-month visit before starting the MERITA treatment. This procedure ensures no bias when assessing the effectiveness of MERITA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient of a Child and Youth Mental Health Center.
* Diagnosis of non-severe mental disorder according to DSM-5 (see exclusion criteria).
* Witness to violence at least in the last two years. A witness to violence is defined at least one of these characteristics (Holden, 2003; Suderman 1999): a) ocular witness of the violence; b) hear violent words or acts when she is in a nearby room; c) living the consequences of the violence without him having seen or heard anything, for example, when he finds that his mother is hurt, that she cries, that she tells him what has happened and that she wants to leave the house, or when he lives the police visit.
* Informed consent of the study signed by the guardian or legal representative.

Exclusion Criteria:

* No signing the informed consent.
* Diagnosis of autism spectrum disorder, active psychotic disorders (schizophrenia, schizophreniform, schizoaffective, brief psychotic disorder, induced psychotic disorder), and severe eating disorder.
* Reason for consultation of forensic evaluation.
* Lack of clear collaboration of adults.
* IQ < 70.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient of a Child and Youth Mental Health Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic symptoms | Baseline
  Children- Adolescent UCLA PTSD Index for DSM-IV (Pynoos et al., 1987). The scale is divided into four dimensions: reexperimentation, behavioral/ cognitive avoidance, cognitive/ mood alterations, and hyperactivation.
Post-traumatic symptoms | Immediately after the intervention
  Children- Adolescent UCLA PTSD Index for DSM-IV (Pynoos et al., 1987). The scale is divided into four dimensions: reexperimentation, behavioral/ cognitive avoidance, cognitive/ mood alterations, and hyperactivation.
Post-traumatic symptoms | 3-month follow-up
  Children- Adolescent UCLA PTSD Index for DSM-IV (Pynoos et al., 1987). The scale is divided into four dimensions: reexperimentation, behavioral/ cognitive avoidance, cognitive/ mood alterations, and hyperactivation.
Post-traumatic symptoms | 6-month follow-up
  Children- Adolescent UCLA PTSD Index for DSM-IV (Pynoos et al., 1987). The scale is divided into four dimensions: reexperimentation, behavioral/ cognitive avoidance, cognitive/ mood alterations, and hyperactivation.
Post-traumatic symptoms | 12-month follow-up
  Children- Adolescent UCLA PTSD Index for DSM-IV (Pynoos et al., 1987). The scale is divided into four dimensions: reexperimentation, behavioral/ cognitive avoidance, cognitive/ mood alterations, and hyperactivation.
Anxiety symptoms | Baseline
  Self-Assessment Questionnaire Anxiety State / Trait in Children -STAIC- by Charles, D. Spielberger, (1982), adapted into Spanish by Seisdedos (1990). It consists of two dimensions: State Anxiety and Trait Anxiety.
Anxiety symptoms | Immediately after the intervention
  Self-Assessment Questionnaire Anxiety State / Trait in Children -STAIC- by Charles, D. Spielberger, (1982), adapted into Spanish by Seisdedos (1990). It consists of two dimensions: State Anxiety and Trait Anxiety.
Anxiety symptoms | 3-month follow-up
  Self-Assessment Questionnaire Anxiety State / Trait in Children -STAIC- by Charles, D. Spielberger, (1982), adapted into Spanish by Seisdedos (1990). It consists of two dimensions: State Anxiety and Trait Anxiety.
Anxiety symptoms | 6-month follow-up
  Self-Assessment Questionnaire Anxiety State / Trait in Children -STAIC- by Charles, D. Spielberger, (1982), adapted into Spanish by Seisdedos (1990). It consists of two dimensions: State Anxiety and Trait Anxiety.
Anxiety symptoms | 12-month follow-up
  Self-Assessment Questionnaire Anxiety State / Trait in Children -STAIC- by Charles, D. Spielberger, (1982), adapted into Spanish by Seisdedos (1990). It consists of two dimensions: State Anxiety and Trait Anxiety.
Depressive symptoms | Baseline
  Childhood Depression Inventory (CDI) (Kovacs, 2004). It contains two subscales: Dysphoria and Negative Self-Esteem.
Depressive symptoms | Immediately after the intervention
  Childhood Depression Inventory (CDI) (Kovacs, 2004). It contains two subscales: Dysphoria and Negative Self-Esteem.
Depressive symptoms | 3-month follow-up
  Childhood Depression Inventory (CDI) (Kovacs, 2004). It contains two subscales: Dysphoria and Negative Self-Esteem.
Depressive symptoms | 6-month follow-up
  Childhood Depression Inventory (CDI) (Kovacs, 2004). It contains two subscales: Dysphoria and Negative Self-Esteem.
Depressive symptoms | 12-month follow-up
  Childhood Depression Inventory (CDI) (Kovacs, 2004). It contains two subscales: Dysphoria and Negative Self-Esteem.
Emotional dysegulation | Baseline
  Scale of difficulties in emotional regulation (DERS) (Gratz and Roemer, 2004) in Spanish. These items are grouped into six subscales: non-acceptance, goals, impulsivity, strategies, awareness, and clarity.
Emotional dysegulation | Immediately after the intervention
  Scale of difficulties in emotional regulation (DERS) (Gratz and Roemer, 2004) in Spanish. These items are grouped into six subscales: non-acceptance, goals, impulsivity, strategies, awareness, and clarity.
Emotional dysegulation | 3-month follow-up
  Scale of difficulties in emotional regulation (DERS) (Gratz and Roemer, 2004) in Spanish. These items are grouped into six subscales: non-acceptance, goals, impulsivity, strategies, awareness, and clarity.
Emotional dysegulation | 6-month follow-up
  Scale of difficulties in emotional regulation (DERS) (Gratz and Roemer, 2004) in Spanish. These items are grouped into six subscales: non-acceptance, goals, impulsivity, strategies, awareness, and clarity.
Emotional dysegulation | 12-month follow-up
  Scale of difficulties in emotional regulation (DERS) (Gratz and Roemer, 2004) in Spanish. These items are grouped into six subscales: non-acceptance, goals, impulsivity, strategies, awareness, and clarity.
Internalizing and externalizing symptoms, prosocial behavior, and interpersonal challenges | Baseline
  Strengths and difficulties questionnaire (SDQ) (Goodman, 1997). It is grouped into five scales: emotional symptoms, behavior problems, hyperactivity/ lack of attention, peer relationship problems, and prosocial behavior.
Internalizing and externalizing symptoms, prosocial behavior, and interpersonal challenges | Immediately after the intervention
  Strengths and difficulties questionnaire (SDQ) (Goodman, 1997). It is grouped into five scales: emotional symptoms, behavior problems, hyperactivity/ lack of attention, peer relationship problems, and prosocial behavior.
Internalizing and externalizing symptoms, prosocial behavior, and interpersonal challenges | 3-month follow-up
  Strengths and difficulties questionnaire (SDQ) (Goodman, 1997). It is grouped into five scales: emotional symptoms, behavior problems, hyperactivity/ lack of attention, peer relationship problems, and prosocial behavior.
Internalizing and externalizing symptoms, prosocial behavior, and interpersonal challenges | 6-month follow-up
  Strengths and difficulties questionnaire (SDQ) (Goodman, 1997). It is grouped into five scales: emotional symptoms, behavior problems, hyperactivity/ lack of attention, peer relationship problems, and prosocial behavior.
Internalizing and externalizing symptoms, prosocial behavior, and interpersonal challenges | 12-month follow-up
  Strengths and difficulties questionnaire (SDQ) (Goodman, 1997). It is grouped into five scales: emotional symptoms, behavior problems, hyperactivity/ lack of attention, peer relationship problems, and prosocial behavior.

SECONDARY OUTCOMES:
Somatic complaints | Baseline
  List of somatic complaints (SCL) (Rieffe et al., 2006; Rieffe et al., 2007) (Górriz, Prat-Gascó, Villanueva and González, 2015).
Somatic complaints | Immediately after the intervention
  List of somatic complaints (SCL) (Rieffe et al., 2006; Rieffe et al., 2007) (Górriz, Prat-Gascó, Villanueva and González, 2015).
Somatic complaints | 3-month follow-up
  List of somatic complaints (SCL) (Rieffe et al., 2006; Rieffe et al., 2007) (Górriz, Prat-Gascó, Villanueva and González, 2015).
Somatic complaints | 6-month follow-up
  List of somatic complaints (SCL) (Rieffe et al., 2006; Rieffe et al., 2007) (Górriz, Prat-Gascó, Villanueva and González, 2015).
Somatic complaints | 12-month follow-up
  List of somatic complaints (SCL) (Rieffe et al., 2006; Rieffe et al., 2007) (Górriz, Prat-Gascó, Villanueva and González, 2015).
Child/adolescents attachment with mother and father | Baseline
  Parental Bonding Instrument (PBI) (Parker, Tupling, and Brown, 1979). It consists of two dimensions: care and overprotection.
Child/adolescents attachment with mother and father | Immediately after the intervention
  Parental Bonding Instrument (PBI) (Parker, Tupling, and Brown, 1979). It consists of two dimensions: care and overprotection.
Child/adolescents attachment with mother and father | 3-month follow-up
  Parental Bonding Instrument (PBI) (Parker, Tupling, and Brown, 1979). It consists of two dimensions: care and overprotection.
Child/adolescents attachment with mother and father | 6-month follow-up
  Parental Bonding Instrument (PBI) (Parker, Tupling, and Brown, 1979). It consists of two dimensions: care and overprotection.
Child/adolescents attachment with mother and father | 12-month follow-up
  Parental Bonding Instrument (PBI) (Parker, Tupling, and Brown, 1979). It consists of two dimensions: care and overprotection.
Family functioning | Baseline
  McMaster Family Assessment Device (FAD) (Epstein, Baldwin, and Bishop, 1983). It contains six dimensions: problem-solving, communication, roles, affective response, emotional involvement, behavioral control, and general family functioning.
Family functioning | Immediately after the intervention
  McMaster Family Assessment Device (FAD) (Epstein, Baldwin, and Bishop, 1983). It contains six dimensions: problem-solving, communication, roles, affective response, emotional involvement, behavioral control, and general family functioning.
Family functioning | 3-month follow-up
  McMaster Family Assessment Device (FAD) (Epstein, Baldwin, and Bishop, 1983). It contains six dimensions: problem-solving, communication, roles, affective response, emotional involvement, behavioral control, and general family functioning.
Family functioning | 6-month follow-up
  McMaster Family Assessment Device (FAD) (Epstein, Baldwin, and Bishop, 1983). It contains six dimensions: problem-solving, communication, roles, affective response, emotional involvement, behavioral control, and general family functioning.
Family functioning | 12-month follow-up
  McMaster Family Assessment Device (FAD) (Epstein, Baldwin, and Bishop, 1983). It contains six dimensions: problem-solving, communication, roles, affective response, emotional involvement, behavioral control, and general family functioning.

OTHER OUTCOMES:
Sociodemographic variables | Baseline
  Sex, age, educational level, number of visits, diagnosis.
Risk factors | Baseline
  Direct abuse, sexual abuse, parental mental disorder, parental alcohol abuse.
Number of attendance at MERITA sessions | Immediately after the intervention
  As a control variable.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Salut Mental Infantojuvenil, Cornellà de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No